CLINICAL TRIAL: NCT06139302
Title: Pharmacokinetics of R-BI 1015550 After Single Oral Doses of BI 1015550 in Japanese Healthy Male Subjects (Open-label, Non-randomised, and Parallel Group Design)
Brief Title: A Study to Test How Different Doses of Nerandomilast (BI 1015550) Are Taken up in the Body of Healthy Japanese Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0038
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Results first posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — BI 1015550

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nerandomilast 9 mg (Experimental): Participants were administered a single film-coated tablet of 9 mg of nerandomilast (Formulation C1), orally with 240 milliliters (mL) of water after an overnight fast of at least 10 hours (h).
  Interventions: Drug: Nerandomilast
- Nerandomilast 18 mg (Experimental): Participants were administered a single film-coated tablet of 18 mg of nerandomilast (Formulation C1), orally with 240 milliliters (mL) of water after an overnight fast of at least 10 hours (h).
  Interventions: Drug: Nerandomilast

INTERVENTIONS:
Drug: Nerandomilast — Participants were administered a single film-coated tablet of nerandomilast (Formulation C1), orally with 240 milliliters (mL) of water after an overnight fast of at least 10 hours (h).
  Other Names: BI 1015550; JASCAYD®

SUMMARY:
The main objectives of this trial are to investigate pharmacokinetics (PK) of R-BI 1015550 in Japanese healthy male subjects following oral administration of two different single BI 1015550 doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR), Respiratory rate (RR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (inclusive)
* Body mass index (BMI) of 18.5 to 25 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR, RR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre(s) of mercury (mmHg), diastolic blood pressure outside the range of 40 to 90 mmHg, or PR outside the range of 40 to 99 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label, non-randomized, and parallel group design study aimed to investigate pharmacokinetics of R-BI 1015550 (nerandomilast) in healthy Japanese male subjects following oral administrations of a single nerandomilast dose of 9 milligrams (mg) or 18 mg.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Nerandomilast 9 mg | Nerandomilast 18 mg
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all subjects who were treated with at least one dose of trial drug. The treatment assignments were determined based on the first treatment the subjects received. The treated set was used for safety analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nerandomilast 9 mg | Nerandomilast 18 mg | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.8 (10.1) | 26.2 (9.6) | 29.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Nerandomilast in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-inf)
Description: Area under the concentration-time curve of nerandomilast in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf) is reported.
Time Frame: Within 3 hours (hrs) before drug intake and at 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 and 144 hrs after drug intake.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): The PKS set included all subjects in the treated set (TS) who provided at least one PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if he contributed only one PK parameter value for one period to the statistical assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanomoles/Liter (h*nmol/L)
Groups:
- Nerandomilast 9 mg: Participants were administered a single film-coated tablet of 9 mg of nerandomilast (Formulation C1), orally with 240 milliliters (mL) of water after an overnight fast of at least 10 hours (hrs).
- Nerandomilast 18 mg: Participants were administered a single film-coated tablet of 18 mg of nerandomilast (Formulation C1), orally with 240 milliliters (mL) of water after an overnight fast of at least 10 hours (hrs).
Arm/Group | Nerandomilast 9 mg | Nerandomilast 18 mg
Number analyzed (Participants) | 6 | 6
hours*nanomoles/Liter (h*nmol/L) | 2070 (13.8) | 3740 (52.8)

2. Primary Outcome: Maximum Measured Concentration (Cmax) of Nerandomilast in Plasma
Description: Maximum measured concentration (Cmax) of nerandomilast in plasma is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles/Liter (nmol/L)
Arm/Group | Nerandomilast 9 mg | Nerandomilast 18 mg
Number analyzed (Participants) | 6 | 6
nanomoles/Liter (nmol/L) | 455 (10.6) | 628 (138)

ADVERSE EVENTS:
Time Frame: Serious adverse events, other adverse events and all-cause mortality: From time of trial drug administration up to 7 days.
Description: Adverse events were reported for the treated set (TS). The treated set included all subjects who were treated with at least one dose of nerandomilast. The treatment assignments were determined based on the first treatment the subjects received. The treated set was used for safety analyses.
Arm/Group | Nerandomilast 9 mg | Nerandomilast 18 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nerandomilast 9 mg (N=6) | Nerandomilast 18 mg (N=6)
Nasopharyngitis (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-08-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT06139302/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT06139302/SAP_001.pdf